CLINICAL TRIAL: NCT03324451
Title: The Effectiveness of Intervention on Insulin Injection in Insulin-naive Patients With Type 2 Diabetes: Application of the Transtheoretical Model
Brief Title: The Effectiveness of Intervention on Insulin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ruey-Hsia Wang, PhD, Professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-E(I)-20150262
Record Dates: First submitted 2017-08-29; First posted 2017-10-27 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Patients with T2DM at a clinic in southern Taiwan are assigned to the intervention arm, whereas patients with T2DM at the endocrinology department of a hospital in northern Taiwan are placed in the control arm. Eligible patients that match the inclusion criteria are recommended by doctors to initiate insulin treatment. Research assistants will explain the objectives of this study to eligible participants. Subsequently, baseline data will be collected from participants by research assistants after the participants sign the consent forms. Afterwards, the participants in the intervention arm will receive the intervention. For the control arm, the participants will receive regular patient education originally administered at the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The arm that receives "TTM Intervention for Insulin Initiation." The intervention contains two parts: (1) individual intervention; (2) insulin injection follow-up management
  Interventions: Behavioral: TTM Intervention for Insulin Initiation
- Control arm (Placebo Comparator): The arm that receives usual care from the hospital that hosts the control arm. Participants in the control arm receives regular patient education.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: TTM Intervention for Insulin Initiation — The intervention contains two parts: (1) individual intervention; (2) insulin injection follow-up management. Different intervention strategies are applied to patients according to their stages of change.
  Arms: Intervention arm
Behavioral: Usual care — Regular patient education on insulin injection at the control arm hospital.
  Arms: Control arm

SUMMARY:
The aim of the study is to assess the effectiveness of an intervention for insulin injection initiation based on the Transtheoretical Model (TTM) for insulin-naïve patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
According to the Transtheoretical Model (TTM) proposed by Prochaska and Diclemente, people will experience different stages of change before the actual behavioral change takes place. Ineffectiveness of intervention to instigate behavioral change is largely due to failure to take into account the stage of change in which individuals are. The TTM suggests that decisional balance, which reflects the relative difference between pros and cons, is important for influencing the stage of change. In order to achieve behavioral change, the perceived pros of changing must be strengthened to outweigh the cons. In addition, individual must be self-convinced that the behavioral change is important for themselves. Furthermore, the process for behavioral change can be provided to facilitate behavioral change in individuals. The theory of TTM has yet been used to improve the behavior of insulin initiation in insulin-naïve patients with T2DM. Thus, this study aims to assess the effectiveness of an intervention for insulin injection initiation based on the TTM in insulin-naïve patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

(1) diagnosed with T2DM for at least half a year; (2) aged 20-70 years old; (3) controlling diabetes only through oral medication, without previous experience in insulin injection; (4) HbA1c≧8.5% as measured more than twice in a year; (5) considered suitable and recommended by the doctor to initiate insulin injection.

Exclusion Criteria:

(1) unable to communicate with language; (2) incapable of self-administering insulin injection due to visual or muscular impairment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Hsia Wang, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Lee's clinic, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 97 | 54
Completed | 65 | 41
Not Completed | 32 | 13

BASELINE CHARACTERISTICS:
Groups:
- Intervention Arm: The arm that receives "TTM Intervention for Insulin Initiation." The intervention contains three parts: (1) individual intervention; (2) insulin injection follow-up management
  TTM Intervention for Insulin Initiation: The intervention contains two parts: (1) individual intervention; (2) insulin injection follow-up management. Different intervention strategies are applied to patients according to their stages of change.
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 97 | 54 | 151
Age, Categorical [Count of Participants; unit: Participants] — Population: some participants were lost
  Participants
    number analyzed (Participants) | 65 | 41 | 106
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 38 | 25 | 63
    >=65 years | 27 | 16 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: some participants were lost follow-up
  years
    number analyzed (Participants) | 65 | 41 | 106
    (all) | 60.91 (14.30) | 60.02 (11.49) | 60.57 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: some participants were lost follow-up
  Participants
    number analyzed (Participants) | 65 | 41 | 106
    Female | 30 | 23 | 53
    Male | 35 | 18 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 97 | 54 | 151

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin (HbA1c) Levels
Description: Collected from blood test to assess the Glycosylated hemoglobin (HbA1c) levels
Time Frame: At baseline and 12 months after the intervention
Measure: Mean (Standard Deviation); unit: percent of glycosylated Hb
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 65 | 41
percent of glycosylated Hb | -1.47 (2.23) | -2.00 (2.29)

2. Secondary Outcome: Change in Diabetes Empowerment Process
Description: A 13-item Chinese version of the Diabetes Empowerment Process Scale was used to assess the perceived level of empowerment by healthcare providers in participants. Each item was rated on a 5-point scale with scores ranging from 0 (strongly disagree) to 4 (strongly agree). The total score range from 13 to 65. A higher score indicated higher perceived patient empowerment.
Time Frame: At baseline and 12 months after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 65 | 41
score on a scale | 0.52 (12.13) | -2.13 (10.99)

3. Secondary Outcome: Change in Diabetes Distress
Description: An 8-item Chinese version of the short-form Problem Areas in Diabetes Scale was used to assess the levels of diabetes distress in participants. The response of each item was rated from 0 (not a problem) to 4 (serious problem). The total score ranged from 8 to 32. A higher score represented severer diabetes distress.
Time Frame: At baseline and 12 months after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 65 | 41
score on a scale | -2.91 (8.16) | -3.63 (6.76)

4. Secondary Outcome: Change in Quality of Life
Description: A 15-item Diabetes-Specific Quality-of-Life Scale was used to assess the subjective appraisal of participants in their perceived degree to which their current health-related aspects in life were affected by emotional suffering, social functioning, adherence to treatment regimen, and diabetic-specific symptoms. Each item was rated from "very much" (0 point) to "not at all" (4 points). The total score ranged from 0 to 60. A higher score indicated better quality of life.
Time Frame: At baseline and 12 months after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 65 | 41
score on a scale | 2.6 (7.51) | 5.45 (10.86)

5. Secondary Outcome: Change in Body Mass Index
Description: Physiological parameter which will be collected from body weight scale and height scale, and will be converted to body mass index (weight (kg)/ height(m) 2
Time Frame: At baseline and 12 months after the intervention
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 65 | 41
Kg/m^2 | 1.06 (1.61) | 0.85 (1.81)

ADVERSE EVENTS:
Time Frame: the adverse event data were collected at 12 months after intervention
Groups:
- TTA Intervention: The intervention contains two parts: (1) individual intervention; (2) insulin injection follow-up management.
- Control Arm: Participants in the control arm receives regular patient education.
Arm/Group | TTA Intervention | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/54
Other Adverse Events (participants affected / at risk) | 0/97 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT03324451/Prot_SAP_000.pdf